CLINICAL TRIAL: NCT07053033
Title: Laser Interstitial Thermal Therapy (LITT) or Surgery and Adjuvant Reirradiation for Recurrent Brain Metastases (LaSAR BeaM)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0377; NCI-2025-04737 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-06-30; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eligible for surgery or LITT-Surveillance (Experimental): Patients will be randomized in a 1:1 manner to close surveillance versus SRS2.
  Interventions: Procedure: Surgery; Procedure: LITT
- Eligible for surgery or LITT-SRS2 (Experimental): Patients will be randomized in a 1:1 manner to close surveillance versus SRS2.
  Interventions: Procedure: Surgery; Procedure: LITT
- Ineligible for surgery or LITT-SRS2 (Experimental): Patients will be randomized in a 1:1 manner to close surveillance versus SRS2.
  Interventions: Procedure: Surgery; Procedure: LITT

INTERVENTIONS:
Procedure: Surgery — Participants will initially undergo craniotomy and surgical resection of lesions or LITT
Procedure: LITT — Participants will undergo 4-core stereotactic biopsy and LITT by experienced neurosurgeons with specific expertise.

SUMMARY:
standard paradigm for management of patients who present with concern for recurrence of brain metastases following initial stereotactic radiosurgery (SRS).

DETAILED DESCRIPTION:
Primary Objective:

To determine whether SRS2 following surgery/LITT for patients with recurrent previously irradiated brain metastases improves time to local recurrence compared to close surveillance following surgery/LITT.

To summarize time to local recurrence for patients with recurrent previously irradiated brain metastases receiving SRS2 due to being ineligible for surgery/LITT.

Secondary Objectives:

To test if the effect of SRS2 versus surveillance after LITT or surgery in patients with recurrent previously irradiated brain metastases is associated with the type of surgical intervention.

To determine whether SRS2 versus close surveillance following surgery/LITT for recurrent previously irradiated brain metastases improves distant brain metastasis-free survival, intracranial progression-free survival, overall progression-free survival, neurologic death rates, and/or overall survival.

To summarize distant brain metastasis-free survival, intracranial progression-free survival, overall progression-free survival, neurologic death rates, and/or overall survival for patients receiving SRS2 alone for recurrent, previously irradiated brain metastases.

To summarize patient-reported outcomes including neurocognitive symptoms, functional independence, and quality of life for patients who receive SRS2 for recurrent, previously irradiated brain metastases.

To summarize radionecrosis and adverse event rates for patients who receive SRS2 following surgery/LITT for recurrent previously irradiated brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Willingness to comply with all study procedures and availability for the duration of the study.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of SRS2, children are excluded from this study.
* Karnofsky performance status ≥ 60.
* Radiographic concern for progression of a solid tumor brain metastasis that has received prior stereotactic radiosurgery ≥ 3 months prior to study enrollment.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as ≥5 mm with MRI scan.
* Have active tumor on pathology from surgery/LITT for this lesion.
* Able to safely undergo MRI imaging.
* Acceptable candidate for SRS2 per treating physician and multidisciplinary conference consensus.
* Have no radiographic evidence of leptomeningeal disease on radiology report or neuro-radiologist review.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria:

* Patients with brain metastases from hematologic malignancies due to significant differences in radiosensitivity and treatment paradigms.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because radiation has the potential for teratogenic or abortifacient effects. All female patients between the onset of menses and 55 years will receive a pregnancy test prior to SRS2 unless the patient presents with an applicable exclusionary factor which may be one of the following:
* Postmenopausal (no menses in greater than or equal to 12 consecutive months).
* History of hysterectomy or bilateral salpingo-oophorectomy.
* Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
* History of bilateral tubal ligation or another surgical sterilization procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Subha Perni, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org